CLINICAL TRIAL: NCT03883789
Title: Defining 'Normal' Liver Function Tests and FibroScan Values in Pregnancies With or Without Liver Disease
Brief Title: Defining 'Normal' Liver Function Tests & FibroScan Values in Pregnancy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: King's College Hospital NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: IRAS 255412
Record Dates: First submitted 2019-02-05; First posted 2019-03-21 (Actual); Last update posted 2019-03-21 (Actual); Status verified 2019-02

CONDITIONS: Pregnancy Disease; Liver Diseases
Keywords: Fibrosis, FibroScan, Pregnancy, Trimesters, Liver disease
MeSH Terms: conditions — Liver Diseases; Fibrosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Normal pregnancies: Participants who have normal uncomplicated pregnancies
  Interventions: Diagnostic Test: FibroScan
- Pregnancies with complications: Participants who undergo pregnancy with liver disease or develop liver disease or other conditions
  Interventions: Diagnostic Test: FibroScan

INTERVENTIONS:
Diagnostic Test: FibroScan — FibroScan will be used to assess liver stiffness

SUMMARY:
The main aim of this single-site prospective study is to use serum liver function tests and FibroScan as assessment tools to measure liver disease in pregnant women with or without liver disease at King's College Hospital. This will be assessed during each trimester of pregnancy. FibroScan will assess liver stiffness in these participants and will be used as a surrogate marker for fibrosis.

DETAILED DESCRIPTION:
Approximately 500 pregnant participants above the age of 16 years will be enrolled into this study, which will occur over an 18-month period (February 2019 to August 2020).

In this prospective cohort study, pregnant participants with or without liver disease will be identified through clinics at King's College Hospital. Participants attending the antenatal, specialist liver-pregnancy clinic and general liver clinics will be given an information leaflet detailing the study. Participants can be interviewed in a clinic room to answer any queries. The participant is then given the option of consenting and participating in the study during that clinic consultation or to contact us at a future date should they need further time for consideration.

Baseline participant details will be collected as well as any preceding liver diagnosis and other comorbidities.

Once consented, the assessment visits will be as follows.

1. Trimester 1 visit (at week 12 booking ultrasound scan):

   - Additional FibroScan after booking scan (ideally 3 hours *fasting will be required before this scan)
2. Trimester 2 visit (at week 20 routine ultrasound scan):

   * Additional FibroScan after ultrasound scan (ideally 3 hours *fasting will be required before this scan)
   * Blood tests to be taken at this point
3. Trimester 3 visit (if occurs, e.g. in participants with diabetes):

   * FibroScan (ideally 3 hours *fasting will be required before this scan)
   * Blood tests (liver function tests)
4. Post-partum visit (if occurs):

   * FibroScan (ideally 3 hours *fasting will be required before this scan)
   * Blood tests (liver function tests)

     * Fasting = nothing to eat or drink (except water)

The participants will be followed up during pregnancy and, if required, for 3 months after pregnancy, as per routine Obstetric care. Delivery, maternal and foetal outcomes will also be documented. This information will come from the participant online medical records.

ELIGIBILITY:
Inclusion Criteria:

* Must be female
* Must be aged 16 years and above and be of childbearing age
* Must be participants attending clinic at King's College Hospital
* Must be in the 1st and 2nd trimester of a pregnancy
* Must be willing and able to provide written informed consent

Exclusion Criteria:

* Non-viable pregnancy
* Pacemaker in situ
* Concurrent and/or recent involvement in other research that is likely to interfere with FibroScan results within last 3 months of study enrolment

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Pregnant women of childbearing age
Study Population: 500 pregnant women above the age of 16 years who will be attending outpatient clinics at King's College Hospital London
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2019-04-01 (Estimated); Primary Completion 2020-10-01 (Estimated); Study Completion 2020-11-01 (Estimated)

PRIMARY OUTCOMES:
The aim of this study is to evaluate the differences in the range of liver stiffness values measured by the 'FibroScan' machine (the measurement tool) between pregnant women with or without liver disease | 18 months
  The objective of this assessment will be to determine normal and abnormal values of liver stiffness within the pregnant population

SECONDARY OUTCOMES:
The normal ranges of liver enzyme levels during pregnancy will be extrapolated from blood sample analysis in the laboratory | 18 months
  Blood tests for liver function tests will be performed at different stages of normal and abnormal pregnancies allowing for analysis to determine normal ranges of values
To evaluate the normal ranges of "Controlled Attenuated Parameter (CAPTM)" values in the pregnant population using FibroScan as the tool to assess this parameter | 18 months
  The FibroScan test will allow the assessment of fat content within the liver in normal and abnormal pregnancies, e.g. those with diabetes
Clinical information in patient notes will be used to evaluate and correlate between different delivery outcomes and FibroScan results in normal and abnormal pregnancies | 18 months
  Various delivery outcomes will be evaluated and correlated against liver stiffness measurement and CAP values (determined by FibroScan), e.g. caesarean section rates
Clinical information in patient notes will be used to evaluate and correlate between different maternal outcomes based on FibroScan results in normal and abnormal pregnancies | 18 months
  Various maternal outcomes will be evaluated and correlated against liver stiffness measurement and CAP values (determined by FibroScan), e.g. hepatic decompensation
Clinical information in patient notes will be used to evaluate and correlate between different foetal outcomes and FibroScan results in normal and abnormal pregnancies | 18 months
  Various foetal outcomes will be evaluated and correlated against liver stiffness measurement and CAP values (determined by FibroScan), e.g. live birth rate

CONTACTS AND LOCATIONS:
Overall Officials: Mussarat N Rahim, MBBSBScMRCP, Principal Investigator — King's College Hospital NHS Trust

IPD SHARING:
Plan to Share IPD: No